CLINICAL TRIAL: NCT04160013
Title: Mitigating ACEs in Pediatric Primary Care: Cohort #2 With 6-24 Month Old Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Seth Scholer, Professor of Pediatrics and Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 171485
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Parenting; Violence; Child Abuse

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Masking Description: No masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discipline education (Experimental): Education about discipline using the Play Nicely program (www.playnicely.org).
  Interventions: Behavioral: Discipline education
- Cavity prevention (Placebo Comparator): Education about cavity prevention using a 2 page handout.
  Interventions: Behavioral: Cavity Prevention

INTERVENTIONS:
Behavioral: Discipline education — Discipline education using the Play Nicely program.
  Arms: Discipline education
Behavioral: Cavity Prevention — Cavity prevention using a 2 page handout.
  Arms: Cavity prevention

SUMMARY:
The aim is to determine if a brief intervention can affect parents' attitudes about physical punishment and other parenting behaviors.

DETAILED DESCRIPTION:
A public health problem that needs to be solved is how to educate more parents about healthy discipline options. The investigators aim to mitigate adverse childhood experiences (ACEs) by integrating evidence-based parent training into pediatric primary care. Some of the most modifiable ACEs are associated with parenting behaviors that can lead to child abuse. The investigators define unhealthy parenting behaviors such as spanking, threatening, yelling, and humiliation. For adults in the original ACEs study, it was exposure to these behaviors that led to the categorization of child abuse/neglect and that were associated with heart disease, obesity, depression, smoking, drug use, violence, and many other problems. This study may help change policy and practice related to mitigating ACEs in primary care. To accomplish this goal, randomized controlled trials are needed to test brief screening tools and evidence-based resources. A population-based approach is needed to reach all parents (i.e. primary prevention). In the study, parents in the intervention group will receive 3 minutes of education about healthy discipline strategies.

ELIGIBILITY:
Inclusion Criteria:

* Parents of 6 month to 2 year old children presenting to the Vanderbilt Pediatric Primary Care Clinic for a well visit or an acute care visit.

Exclusion Criteria:

* Parents who do not speak and read English, Spanish, or Arabic. The interventions are only available in English, Spanish, and Arabic.

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 533 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2019-01-19 (Actual)

PRIMARY OUTCOMES:
Attitudes toward spanking | 3-6 months post-enrollment.
  A 10 item scale that assesses parents' attitudes about corporal punishment. The minimum value is 10 and the maximum value is 70. Higher scores indicate a higher likelihood of using spanking.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States